CLINICAL TRIAL: NCT05692323
Title: A Supervised Prehabilitation Program for Patients With Pancreatic Cancer
Acronym: PREHAB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Philip Chang, Sponsor-Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2021-18-CHANG-PREHAB
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pancreas Cancer
Keywords: Exercise; Prehabilitation
MeSH Terms: conditions — Pancreatic Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supervised Prehabilitation Exercise Program (Experimental)
  Interventions: Other: PREHAB

INTERVENTIONS:
Other: PREHAB — 6-week supervised PREHAB program. Each week of the program consists of 3 x 1 hour supervised training sessions made up of moderate intensity aerobic training and resistance training. In addition to the supervised sessions, patients will be instructed to accumulate a total of 150 minutes per week of moderate aerobic training at home which is measured by a wrist worn FitBit device.

SUMMARY:
The purpose of this study is to assess the use of an exercise program in people with pancreatic cancer.

DETAILED DESCRIPTION:
Attendance to exercise sessions as well as impacts on healthcare utilization, muscle mass, quality of life, physical activity, and post-operative outcomes when applicable will be monitored.

Study participants will participant in a supervised, in-person exercise program 3 times per week for 6 weeks. Participants will receive a Fitbit to be worn continuously during the study and complete surveys and exercise tests at specified timepoints (Baseline, Post-Intervention Evaluation and 3-Month Follow Up).

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cancer diagnosis (any stage)
* Age ≥ 18 years
* Independent ambulation and activities of daily living (Discretion of referring/ treating oncologist)
* Godin-Shephard Leisure-Time Physical Activity Questionnaire score of ≤ 23
* Physically able to complete functional assessments including 6-minute walk test, hand grip strength, short performance physical battery and performance metrics
* Answers no to all questions on PAR-Q OR is cleared to participate by their treating oncologist
* Ability to read, write and understand English
* Written informed consent obtained from subject and ability for subjects to comply with the requirements of the study

Inclusion criteria for remote monitoring of physical activity (Fitbit) and online Pain portal only (failure to meet inclusion criterion below should not preclude subjects from participating in main study):

* Access to a smart device capable of Fitbit syncing and accessing the online Pain portal (www.painguide.com)

Exclusion Criteria:

* Has undergone or plans to undergo resection surgery prior to projected completion of PREHAB exercise intervention
* Current pregnancy

Exclusion criteria for remote monitoring component of the study with Fitbit only (failure to meet exclusion criterion below should not preclude the subject from participating in main study):

* Using a pacemaker, implantable cardiac defibrillator, neurostimulator, cochlear implants (removable hearing aids permitted), or other electronic medical equipment, unless the PI deems study participation safe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
PREHAB Program feasibility will be measured by tracking participant attendance at PREHAB sessions. PREHAB will be considered feasible if 50% of participants attend at least 60% of scheduled sessions. | From Baseline to 3 Months
  PREHAB session feasibility is defined as at least 50% of participants attending at least 60% of scheduled sessions

SECONDARY OUTCOMES:
PREHAB Program safety will be assessed through the reporting of unanticipated problems from the baseline visit through to the 3 Month visit. | From Baseline to 3 Months
  PREHAB program safety will be evaluated by monitoring unanticipated problems involving risk to subjects or others (UPIRSO).

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chang, DO, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No